CLINICAL TRIAL: NCT02046707
Title: Evaluation of the Effects of Eccentric Muscle Training Versus Conventional Concentric Training in Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CASILLAS Fondation Av 2008
Record Dates: First submitted 2014-01-20; First posted 2014-01-28 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Chronic Heart Failure; Reconditioning to Effort

ARMS (2):
- Patients with chronic heart failure (Experimental)
  Interventions: Other: initial evaluation; Other: Period of cardiac rehabilitation; Other: final evaluation
- Controls (Other)
  Interventions: Other: Concentric and eccentric exercise sessions

INTERVENTIONS:
Other: initial evaluation
  Arms: Patients with chronic heart failure
Other: Period of cardiac rehabilitation
  Arms: Patients with chronic heart failure
Other: final evaluation
  Arms: Patients with chronic heart failure
Other: Concentric and eccentric exercise sessions
  Arms: Controls

SUMMARY:
This is a single-centre open randomized parallel-group study. Patients will be selected at random to be included in group 1: eccentric rehabilitation or group 2: conventional rehabilitation.

In addition, a group of healthy volunteers aged between 20 and 85 years will also be recruited. This group will make it possible to evaluate, during the two exercise sessions, mechanisms of adaptation linked to eccentric exercise vs concentric exercise.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Patients who have provided written informed consent
* Patients with national health insurance cover
* Men or women aged between 45 and 85 years with stabilized chronic heart failure (ischemic or dilated cardiopathy) for at least one month, New York Heart Association stage> 2.
* Echocardiographic left ventricular ejection fraction (Simpson method) < 45% OR N-terminal-ProBNP > 3 x upper limit of normal* (*= 125pg/ml for the CHU laboratory).
* First period of rehabilitation for chronic heart failure.

Healthy volunteers:

* Subjects who have provided written informed consent
* Subjects with national health insurance cover
* Men or women aged between 18 and 85 years.

Exclusion Criteria:

Patients:

* persons without national health insurance cover
* Severe obstructive cardiopathy,
* severe aortic valve stenosis,
* severe progressive heart rhythm or conduction disorders not corrected with a pacemaker, discovered at the initial effort test
* intra-cavitary thrombus,
* severe pulmonary artery hypertension (systolic pulmonary arterial hypertension >70mmHg),
* recent history of venous trombo-embolism (last 3 months),
* impaired executive function making it impossible to understand and follow reconditioning programme (Mini Mental Test < 24),
* heart transplant,
* associated medical disorders that could predominately impair functional capacity compared with the chronic heart failure (examples: respiratory insufficiency, non-stabilized metabolic disorders such as progressive kidney failure, severe asthenia related to a severe non-stabilized disorder such as neoplasia, systemic disease…).

associated chronic motor deficit of a neurological origin (example: sequelae of a cerebrovascular accident), an osteo-articular origin (example: impairment due to Rheumatoid arthritis), of a peripheral vascular disease (example: peripheral artery disease, venous disease, lymphedema) will not be included in the exclusion criteria provided thay are compatible with the level of physical ability defined in the inclusion criteria. The presence of an implantable pacemaker and/or defibrillator will not be an exclusion criterion

Healthy volunteers:

* persons without national health insurance cover
* Any organic disorder whatever its nature (cardiac, respiratory, neurological, orthopedic, …) that could affect adaptation to effort or is a contra-indication for physical activity.

Ages: 45 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-08-29 (Actual); Primary Completion 2015-03-23 (Actual)

PRIMARY OUTCOMES:
Evolution of performance in the 6-minute walk test between the initial assessment and the final assessment of a reconditioning programme | 12 weeks

SECONDARY OUTCOMES:
Evolution of functional and physiological capacities and tolerance criteria | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France